CLINICAL TRIAL: NCT05803265
Title: Prevalence of Children Witnessed Violence Evaluated in a Pediatric Emergency Department
Brief Title: Children Witnessed Violence Evaluated in a Pediatric ED
Status: Completed | Type: Observational
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Sponsor
Other Study IDs: RC 14/19
Record Dates: First submitted 2023-03-24; First posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Violence, Domestic; Intimate Partner Violence
Keywords: Witnessed violence; Intimate partner violence; Woman Abusive Screening Tool; Pediatric emergency department

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Witnessed violence is a form of child abuse with detrimental effects on child wellbeing and development, whose recognition relies on the assessment of their mother exposure to intimate partner violence (IPV). The aim of this cross-sectional study is to assess the frequency of witnessed violence in a population of children attending a pediatric emergency department (ED) in Italy, by searching for IPV in their mother, and to define the characteristics of the mother-child dyads.

DETAILED DESCRIPTION:
Witnessed violence is a form of child abuse, consisting of the child experience of any kind of maltreatment against his/her parents/caregivers/family members, and can be either direct (if the maltreatment takes place in the child presence) or indirect (if the child is aware of the maltreatment and perceives its acute/chronic, physical/psychological effects). The recognition of children witnessed violence requires the previous assessment of their mothers' exposure to intimate partner violence (IPV), defined by the World Health Organization (WHO) as a "behavior within an intimate relationship that causes physical, sexual, or psychological harm, including acts of physical aggression, sexual coercion, psychological abuse and controlling behaviors" committed by a current or former partner. According to the WHO reports, one in three women is subjected to IPV, and it has been estimated that among children living in households where IPV takes place, 85% are direct witnesses to violence, and up to one half undergo direct forms of abuse, mostly by the father or any other male family member. Exposure to IPV not only has deleterious effects on the child wellbeing, and cognitive and socio-emotional development, but it also negatively affects behaviors and relationships into adulthood: boys and girls who experience household violence against their mother are at increased risk of perpetuating aggressive behaviors and being victims of domestic violence later in their own lives, respectively, engaging in the so-called intergenerational perpetuation of violence. While the WHO currently recommends screening for IPV during pregnancy, no agreement exists on the appropriateness of routine assessments of postpartum IPV. Nevertheless, on the ground of the detrimental effects of IPV on children, the American Academy of Pediatrics advocated for IPV screening in pediatric settings, endorsing the abuse of women as a pediatric issue. Healthcare professionals are generally in a privileged position to investigate IPV; the emergency department (ED) represents an ideal setting to detect abuse and take actions against it, providing a unique opportunity to involve the mother-child dyads in research surveys, in accordance with the international guidelines on research on violence against women and children. The aim of this study is to assess the frequency of witnessed violence in a population of children attending a pediatric emergency department (ED) in Italy, by searching for IPV in their mother, and to define the characteristics of the mother-child dyads.

ELIGIBILITY:
Inclusion Criteria:

* children aged 0 to 17 years
* attending the pediatric ED (undergoing clinical observation within the ED and/or admission to the ward )
* presence of their mothers

Exclusion Criteria:

* inability of the mother to fill in the questionnaire (due to either language barrier or inability to leave the child behind for a while)
* impossibility to take the mother aside from her partner

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Mother-child dyads attending a pediatric Emergency Department in Italy
Sampling Method: Non-Probability Sample
Enrollment: 212 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
To evaluate the prevalence of children witnessed violence | Within 6 hours of ED admission
  Mothers of children attending a pediatric ED will receive a questionnaire, which will include the validate italian version of Woman Abuse Screening Tool (WAST), a questionnaire assessing women's physical, psychological, and sexual abuse by their partner in the last 12 months. It comprises eight questions, each with three possible answers, graded from 0 (never) to 2 (often): an overall score of 4 or above suggests women abuse by their partner.

SECONDARY OUTCOMES:
To define the demographical and clinical characteristics of the mother-child dyads enrolled | Within 6 hours of ED admission
  Mothers of children attending a pediatric ED will receive a questionnaire which will include questions about their baseline data and health.

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Germani, MD, Principal Investigator — IRCCS materno infantile Burlo Garofolo
Locations (1):
- IRCCS Burlo Garofolo, Trieste, Italy